CLINICAL TRIAL: NCT04041440
Title: Customized Auditory Brain Training for Children With Hearing Loss
Brief Title: Speech Recognition Training in Children With Hearing Loss
Acronym: ChAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201602007
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss
Keywords: Auditory training; Children with hearing loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Within subjects A1 - A2 - B1 - B2 design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auditory Training (Experimental): Pre- and post assessments of auditory training intervention
  Interventions: Behavioral: clEAR auditory training

INTERVENTIONS:
Behavioral: clEAR auditory training — Children play auditory brain training computer games

SUMMARY:
clEAR's auditory brain training has been shown to be effective in improving childrens' abilities to recognize the speech of generic talkers in a laboratory setting. In the proposed research, the researchers will build upon these results and assess the extent to which auditory brain training delivered via the web enhances children's abilities to recognize the speech of a potential classroom teacher and diminishes their communication challenges that are associated with significant hearing loss. First, investigators will conduct focus groups with children who have undergone training with the research version of clEAR's pediatric games, then they will recode the games from LabView to Java Script, making changes in the games in response to the focus group comments, and finally, they will collect data from 20 children to assess whether web-based auditory brain training improves their abilities to recognize the speech of their (hypothetical) upcoming school year's classroom teacher.

DETAILED DESCRIPTION:
Imagine that someday, children with hearing loss can prepare for an upcoming school year by playing computer games with their new teacher's voice throughout the summer. Then, on the first day of class, children would have that "Oprah Winfrey effect", the sense that they know the teacher. Children would be able to recognize their teacher's voice much better than they would have otherwise, and importantly, they would experience less anxiety because of the talker familiarity effect. clEAR is making that "someday" a reality today. clEAR has created a new web-based clinical tool for audiologists and teachers to provide customized auditory brain training to their patients (www.clearforears.com). Auditory brain training includes traditional analytic and synthetic training as well as training to develop those auditory cognitive skills that are necessary to decode spoken language regardless of the content (i.e., auditory working memory, auditory attention, and auditory processing speed). The centerpiece of the clEAR website is a set of auditory brain training games that patients play, with oversight and coaching from their hearing healthcare provider or from one of clEAR's inhouse audiologists. Currently, clEAR caters to adult patients, and the games require some reading ability and a vocabulary that includes the most common words of the English language (N=800 words). clEAR has been enrolling paying adult subscribers since May of 2017. In the laboratory, a research version of pediatric games is being tested. The pediatric games are "childfriendly" and require only a limited vocabulary and no reading skills. In this Phase 1, the investigators will first conduct focus groups with 10 children who have undergone training with the research version of clEAR's pediatric games, then they will recode the games from LabView to Java Script, making changes in the games in response to the focus group comments, and finally, they will collect data from 20 children to assess whether web-based auditory brain training improves their abilities to recognize the speech of their (hypothetical) upcoming school year's classroom teacher. The experimental design will be a within-subjects A1-A2-B1-B2 design, where children will serve as their own controls. Participants will be tested two times before training with a one-week interval separating the test sessions (A1 and A2), to establish a baseline performance, and then immediately after training (B1) to establish immediate gains and three weeks later to assess whether gains begin to decline following training (B2). All testing and training will occur during the summer so the experimental results will not be confounded by benefits possibly accrued through school-related activities. Children will complete a total of 16 hours of training and will follow the same schedule (i.e., play the games in a prescribed order and for a set amount of time each). Outcome measures will come from a comprehensive speech perception test battery, questionnaires, and from data collected during training and stored on the children's training tablets. In Phase II, the pediatric games will be transferred to the clEAR website and develop their commercial potential.

ELIGIBILITY:
Inclusion Criteria:

* Children with moderate to severe hearing loss.

Exclusion Criteria:

* Must be native English speakers

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris A Cardinal, PhD, Principal Investigator — clEAR: Customized Hearing
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Only descriptive data will be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- Focus Groups: Two groups of children participated in focus groups (N=7 and N=5). Results of subjective questions and focused conversations from the focus groups were used to update and modify the clEAR games to make them more fun and engaging.
- Auditory Training Group: One group of children participated in auditory training (N=20 completed the protocol, 22 were consented). Results of objective pre- and post-training assessments from the training group were compared to evaluate the effectiveness of the games.
Period: Overall Study
Arm/Group | Focus Groups | Auditory Training Group
Started | 12 | 22
Completed | 12 | 20
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Auditory Training: Pre- and post assessments of auditory training intervention
  clEAR auditory training: Children play auditory brain training computer gamesFocus
- Focus Group: Two focus groups
  Focus groups to collect feedback on current version of games
- Total: Total of all reporting groups
Arm/Group | Auditory Training | Focus Group | Total
Number analyzed (Participants) | 22 | 12 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (1.3) | 7.28 (1.37) | 9.45 (2.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 8 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 19 | 8 | 27
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 12 | 5 | 17
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 12 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Words Identified Before and After Training
Description: The measure is percent of 50 common words correctly identified. Words were presented through the application and responses were recorded and scored by the audiologist administering the test.
Time Frame: Before and after the four week training period
Population: Data are for children with hearing loss who participated in the auditory training part of the study. One participant in the auditory training group was unable to complete the assessments before and after the training because their speech perception ability was below the level of the assessment material. They were allowed to continue the training part of the study to see if they could still be helped by the training. Outcome measures were not collected from the Focus group.
Measure: Mean (Standard Deviation); unit: percentage of words presented
Groups:
- Auditory Training Group: Children playing auditory brain training computer games
Arm/Group | Auditory Training Group
Number analyzed (Participants) | 19
percentage of words presented
  Pre-Training Scores | 49.7 (13.2)
  Post-Training Scores | 55.7 (17.6)

2. Secondary Outcome: Processing Speed
Description: How quickly, in milliseconds, a word can be discriminated from a competitor
Time Frame: over course of 4 weeks
Population: Data were not collected as the protocol was revised to include only testing that could be conducted remotely. This type of cognitive task requires monitored testing procedures.
Groups:
- Auditory Training Group: Children with hearing impairment playing auditory brain training computer games
Arm/Group | Auditory Training Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Working Memory
Description: Number of words remembered from a list of words presented sequentially
Time Frame: over course of 4 weeks
Population: as for outcome 2
Arm/Group | Auditory Training Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Subjective Assessment of clEAR Games on a 7-Point Scale
Description: clEAR Questionnaire is given to provide researchers feedback and suggestions about the clEAR games from the child's perspective. The questionnaire used 7-point Likert scales, yes-no questions, open ended questions. Average scores across all of the Likert scale questions are reported here because they are quantifiable. Here are the questions analyzed.
  1. How much did you like the home training program?
  2. Do you think playing the games improved your speech discrimination abilities? (how well you understand speech)
  3. Do you think playing the games improved your confidence in conversation?
  4. Did you enjoy playing the games in your home?
  5. How likely would you be to tell your friends who have hearing loss about this program?
  Participants were asked to respond to each item using this scale:
  (very little) 1 2 3 4 5 6 7 (very much)
Time Frame: Measured once, after the four week training period
Population: Data are for children with hearing loss who participated in the auditory training part of the study. Outcome measures were not collected from the Focus Group.
Measure: Mean (Standard Deviation); unit: Units on a 7-point scale
Groups:
- Auditory Training Group: Children that played the auditory brain training computer games
Arm/Group | Auditory Training Group
Number analyzed (Participants) | 20
Units on a 7-point scale | 5.25 (1.41)

ADVERSE EVENTS:
Time Frame: Three Months
Description: No adverse events were anticipated.
Arm/Group | Focus Groups | Auditory Training Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/22
Other Adverse Events (participants affected / at risk) | 0/12 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT04041440/Prot_SAP_000.pdf
  • Informed Consent Form: Consent Information Sheet for Participation in AT (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT04041440/ICF_001.pdf
  • Informed Consent Form: Informed Consent for Focus group (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT04041440/ICF_002.pdf